CLINICAL TRIAL: NCT06942520
Title: A Randomized, Open Label, Controlled, Phase 2 Clinical Study to Evaluate the Efficacy and Safety of RGX-314 AAV Gene Therapy Administered Via Subretinal Delivery in Participants With Center Involved Diabetic Macular Edema
Brief Title: Phase 2 Trial of RGX-314 in Adults With Center Involved - Diabetic Macular Edema (CI - DME)
Acronym: ELAAVATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Eye Associates (Other)
Collaborators: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEA1979
Record Dates: First submitted 2024-12-03; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; gene therapy
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- RGX-314 Treatment Arm (Dose 1) (Experimental): Genetic: RGX-314 Dose 1
  - AAV8 vector containing a transgene for anti-VEGF fab (Dose 1)
  Interventions: Genetic: RGX-314 Dose 1
- Treatment Arm (Dose 2) (Experimental): Genetic: RGX-314 Dose 2
  -AAV8 vector containing a transgene for anti-VEGF fab (Dose 2)
  Interventions: Genetic: RGX-314 Dose 2
- Aflibercept Treatment Arm (Active Comparator): Biological: Aflibercept IVT
  * Commercially available Active Comparator
  * Other Names: Eylea
  Interventions: Biological: Aflibercept (2.0 mg)

INTERVENTIONS:
Genetic: RGX-314 Dose 1 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 1)
  Arms: RGX-314 Treatment Arm (Dose 1)
Genetic: RGX-314 Dose 2 — AAV8 vector containing a transgene for anti-VEGF fab (Dose 2)
  Arms: Treatment Arm (Dose 2)
Biological: Aflibercept (2.0 mg) — Commercially available Active Comparator
  Arms: Aflibercept Treatment Arm

SUMMARY:
Phase 2 open label, randomized, active controlled, dose-ranging trial in adults with Center Involved - Diabetic Macular Edema (CI - DME)

DETAILED DESCRIPTION:
This Phase 2 trial is an open label, randomized, active controlled, dose-ranging trial to allow for preliminary safety and efficacy data on subretinal (SR) delivery of RGX-314 in participants with CI - DME

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II diabetes mellitus with center involving diabetic macular edema with previous treatment
* HbA1c ≤12%
* BCVA in study eye 78 to 25 ETDRS letters (~20/32 to 20/320) at screening
* Decreased visual acuity attributable primarily due to CI - DME
* Demonstrate clinical response to aflibercept injection in the study eye
* Provide written informed consent

Exclusion Criteria:

* Women of childbearing potential
* Neovascularization in the study eye from a cause other than DR
* Evidence in the study eye of optic nerve pallor on clinical examination
* History of pan retinal photocoagulation in the study eye
* Any concurrent ocular condition in the study eye other than CI-DME that could require surgical intervention within 6 months or any condition in the study eye that may increase the risk to the participant, require either medical or surgical intervention during the study to prevent or treat vision loss, or interfere with the study procedures or assessments
* Presence of an implant in the study eye at screening (excluding intraocular lens)
* Any condition in the investigator's opinion that could limit VA improvement in the study eye
* Active or history of glaucoma, steroid response, or ocular hypertension
* Any prior intravitreal steroid injection in the study eye within 6 months prior to screening, administration in the study eye of Ozudrex® within 12 months prior to screening, or administration in the study eye if Iluven® within 36 months prior to screening
* Diabetic macular edema diagnosis ≥ 7 years
* History of chronic renal failure requiring dialysis or kidney transplant
* Participation in any other gene therapy study or receipt of any investigational product within 30 days prior to enrollment or 5 half-lives of the investigational product, whichever is longer, or any plans to use an investigational product within 6 months following enrollment

Note: Other inclusion/exclusion criteria apply

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA in the study eye at Week 52 | 52 Weeks
  To evaluate the effect of RGX-314 on BCVA at Week 52

SECONDARY OUTCOMES:
Mean change from baseline in BCVA in the study eye over time | 52 Weeks
  To evaluate the effect of RGX-314 on BCVA over time
Proportion of participants with BCVA of 20/40 or better (ETDRS ≥ 69 letters) in the study eye over time | 52 Weeks
  To evaluate the effect of RGX-314 on BCVA over time
Mean change from baseline in central subfield thickness (CST) in the study at week 52 | 52 Weeks
  To evaluate the effect of RGX-314 on anatomic outcomes and CST (as determined by SD OCT measurement) at Week 52
Mean change from baseline in CST in the study eye on SD-OCT at Week 26 and Week 52 | 52 Weeks
  To evaluate the effect of RGX-314 on anatomic outcomes and CST (as determined by SD OCT measurement) at Week 52
Proportion of participants with an absence of CI-DME in the study eye at Week 26 and Week 52 | 52 Weeks
  To evaluate the effect of RGX-314 on anatomic outcomes and CST (as determined by SD OCT measurement) at Week 52
Proportion of participants achieving a 2-step or greater improvement or any improvement (a 1-step or greater improvement) in DR in the study eye by ETDRS DRSS on 4 widefield digital stereoscopic fundus photography at Week 52 | 52 Weeks
  To evaluate the effect of RGX-314 on DR by the ETDRS DRSS at Week 52
Incidences of overall and ocular adverse events (AEs) | 52 Weeks
  To assess the safety and tolerability of RGX-314
Proportion of participants requiring any additional intervention for ocular diabetic complications to Week 52 | 52 Weeks
  To evaluate the need for additional standard of care intervention due to ocular diabetic complications
Proportion of participants with any sight-threatening ocular diabetic complications to Week 52 | 52 Weeks
  To evaluate the need for additional standard of care intervention due to ocular diabetic complications
Proportion of participants developing ocular diabetic complications requiring treatment per standard of care (anti-VEGF treatment, steroid treatment, pan retinal photocoagulation, laser, or surgery) through Week 52 | 52 Weeks
  To evaluate the need for additional standard of care intervention due to ocular diabetic complications
Proportion of participants developing ocular diabetic complications (e.g., neovascularization due to DR) requiring treatment per standard of care (pan retinal photocoagulation or anti-VEGF treatment) through Week 52 | 52 Weeks
  To evaluate the need for additional standard of care intervention due to ocular diabetic complications
Proportion of participants developing ocular diabetic complications (e.g., retinal detachments) requiring surgical intervention per standard of care through Week 52 | 52 Weeks
  To evaluate the need for additional standard of care intervention due to ocular diabetic complications
Aqueous RGX-314 transgene (TP) concentration at assessed time points | 52 Weeks
  To measure aqueous RGX-314 TP concentrations
Proportion of participants with visual stability in the study eye from baseline to Week 52 | 52 Weeks
  To evaluate the effect of RGX-314 on vision outcomes
Proportion of participants with vision gain or vision loss ≥ to 5, 10, or 15 ETDRS letters in the study eye from baseline to Week 52 | 52 Weeks
  To evaluate the effect of RGX-314 on vision outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Sierra Eye Associates, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided